CLINICAL TRIAL: NCT04070274
Title: A New Surgery Platform for Calcaneal Surgery: a Clinical Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhuan Zhang, Principal Investigator, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20190810
Record Dates: First submitted 2019-08-15; First posted 2019-08-28 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Calcaneus Fracture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New surgery platform for calcaneal surgery (Experimental): The lateral position surgical platform for calcaneus surgery is designed with a bottom board, mats in front and at back of calf and thigh, and two sizes of cover plates, using "tunnel" principle according to physiological curve of lower limbs.
  Interventions: Procedure: different types of surgery platforms
- Traditional lateral platform (Experimental): The traditional lateral position makes the surgery platform "bread-shaped arch" surface by using medical mats and putting lower limbs superimpose on each other
  Interventions: Procedure: different types of surgery platforms

INTERVENTIONS:
Procedure: different types of surgery platforms — 58 patients with lateral calcaneus surgeries are divided into the control group of 29 patients and the experimental group with 29 patients. The traditional lateral method and calcaneus lateral surgery platforms are separately applied in the groups.

SUMMARY:
Purpose: Study on the method of lateral nursing and surgical operating tables optimization in the calcaneal surgery.

Method:Design combined surgical operating tables grouped according to the time of clinical application.58 patients with lateral calcaneus surgeries are divided into the control group of 29 patients and the experimental group with 29 patients. The traditional lateral method and calcaneus lateral surgery platforms are separately applied to compare the sliding of the affected limb during a surgery, the stability of the position, the difference of the surgical instruments fall and the satisfaction of the medical staff.Moreover,30 healthy volunteers are selected to experience the comfort level of the two placement methods.

ELIGIBILITY:
Inclusion Criteria:

* Ages ranged from 18 to 82.
* ASA Ⅰ or Ⅱ level.

Exclusion Criteria:

* Limited body activity and extremely severe cardiovascular diseases.
* Unwilling to cooperate.
* Mental illness and coagulopathy

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
The sliding frequency of the affected limb during a surgery with two methods | Intraoperative
  More or fewer times
The time patients'surgical position can last for in a surgery. | Intraoperative
  Necessary position stability is significant.For intraoperative fluoroscopy,surgeons need to keep the injured feet a fixing steady position with the help of different platforms.So,time the steady position can last for is recorded by the investigator separately.
The frequency of the surgical instruments fall with different methods | Intraoperative
  More or fewer times
The whole satisfaction level of the patients and medical staffs | From the beginning of operation till 1 days postoperative
  Patients and medical staffs are asked for feelings about the utilization of the new surgical platform.Mark 0 is extreme poor.Mark 10 is very perfect,and the numbers between them are comments of varying degrees.

SECONDARY OUTCOMES:
Extra possible adverse effects due to the new surgical platform | From the beginning of operation till 24 hours postoperative
  Check adverse effects on the basis of influences on respiratory or circulatory systems and damages on patients' nerves or skin.